CLINICAL TRIAL: NCT02630862
Title: Oxidative Stress and Oxysterols Profiling in Patients With Carotid Revascularization: Effect of Antithrombotic Treatment
Brief Title: Oxidative Stress and Oxysterols Profiling in Patients With Carotid Revascularization
Acronym: ICAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Civic Hospital, Italy (Other)
Responsible Party: Principal Investigator, Luigi Iuliano, Associate Professor of Internal Medicine, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IULIANO_Carotids
Record Dates: First submitted 2015-05-26; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Carotid Stenosis; Cardiovascular Disease; Atherosclerosis; Stroke
Keywords: oxidative stress; atherosclerosis; carotid stenosis; oxysterols; vitamin E; lipid peroxidation; antioxidants; aspirin; dipyridamole
MeSH Terms: conditions — Carotid Stenosis; Cardiovascular Diseases; Atherosclerosis; Stroke | interventions — Aspirin; Dipyridamole; Aspirin, Dipyridamole Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Active Comparator): acetylsalcylic acid 100 mg per day give orally for six months, starting the day of carotid endoartherectomy
  Interventions: Drug: Aspirin
- aspirin plus dipyridamole (Active Comparator): acetylsalicylic acid 25 mg plus dipyridamole extended release 200 mg, combined in a capsule, per day starting the day of carotid endoartherectomy
  Interventions: Drug: aspirin plus dipyridamole

INTERVENTIONS:
Drug: Aspirin — Aspirin is a standard and guidelines supported therapy for patients undergoing carotid endoarterectomy as secondary prevention measure of cardiovascular risk
  Other Names: Cardioaspirin, 100 mg; acetylsalicylic acid, 100 mg
  Arms: aspirin
Drug: aspirin plus dipyridamole — the combination of aspirin plus dipyridamole is approved to lower the risk of stroke in people who have had a transient ischemic attack or stroke
  Other Names: aspirin 25 mg plus dipyridamole extended release 200 mg; aggrenox
  Arms: aspirin plus dipyridamole

SUMMARY:
The combination of aspirin and dipyridamole, two antiplatelet drugs, is approved in Italy for the secondary prevention of cerebral embolism in patients with carotid atherosclerosis.

Besides antiplatelet activity, Dipyridamole has additional pharmacological action, including vasodilation and antioxidant properties.

A role for oxidative stress has been suggested in acute cerebrovascular disease. In this study the investigators want to test the in vivo antioxidant activity of dipyridamole in patients who are candidate to take the drug under approved conditions of the Italian Drug Regulation Agency, i.e. secondary prevention of TIA/Stroke in patinets with carotid stenosis (>= 70%).

To test the hypothesis that dipyridamole acts as antioxidant in vivo, oxysterols (products of cholesterol autoxidation) and vitamin E are measured in plasma before and after 6 months therapy after carotid endoarterectomy. Since dipyridamole is approved as combination preparation with aspirin, a control group of patients taking aspirin alone is enrolled.

Outcome measures: plasma biomarkers (oxysterols and vitamin E) change at two time points: baseline and 6-months therapy.

DETAILED DESCRIPTION:
Dipyridamole has been shown to act as potent antioxidant in vitro. The aim of the present study is to analyze if dipyridamole retains the antioxidant in vivo in man.

The investigators identified a clinical setting where dipyridamole is approved for clinical use, i.e. secondary prevention of stroke, to test the hypothesis that dipyridamole given orally could affect circulating markers of oxidative stress, in particular reduction in oxysterols (autoxidation products of cholesterol) and increase in vitamin E concentration.

Methods. Two arms are included in the study: a) dipyridamole plus aspirin (in Italy the use of dipyridamole is approved in combination with aspirin); b) aspirin alone as comparison arm. Patients eligible for endoarterectomy for the presence of carotid stenosis >= 70% are randomized in the two arms. The study is open labeled for the patient and clinical investigators who have in charge the patinets . The study is blinded for the technicians performing biomarker assessment and investigators responsible for data analysis.

Blood is taken at baseline (before surgery) and after six months of treatment. Oxysterol profiling and vitamin E are measured by isotope dilution gas chromatography and mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid atherosclerosis eligible for carotid endoarterectomy (stenosis >= 70%) with previous TIA or Stroke

Exclusion Criteria:

* Congestive heart failure, chronic liver disease, chronic kidney disease (GFR < 60%), cancer, use of antioxidant supplements in the previous 3 months, autoimmune diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Level of oxysterol measured by isotope dilution gas chromatography-mass spectrometry | 6-months
  Oxysterols are used here as markers of oxidative stress, i.e. increased oxidative stress is refected by increased oxysterols levels
Level of alpha- and gamma-tocopherol (vitamin E isomers) by isotope dilution gas chromatography-mass spectrometry | 6-months
  Increased oxidative stress is expected to reduce the levels of of vitamin E isomers by consumption

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Bertoletti, M.D., Principal Investigator — Goretti Hospital, Latina
Locations (1):
- Civic Hospital, Vascular Surgery Unit, Latina, LT, Italy